CLINICAL TRIAL: NCT05951933
Title: Effectiveness of Transcranial Electrical Stimulation in the Functional Recovery of Subjects with Subacromial Pain Syndrome: Randomized Clinical Trial.
Brief Title: Transcranial Electrical Stimulation in Subacromial Pain Syndrome
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Marta Aguilar, Principal investigator, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: UnVa
Record Dates: First submitted 2023-06-29; First posted 2023-07-19 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2024-05

CONDITIONS: Subacromial Pain Syndrome
Keywords: Physiotherapy; Strenghtening; Conservative treatment; Transcranial direct electrical stimulation; Therapeutic exercise; Pain; Functionality; Quality of life; Mucle Strenght; Range of movement; Proprioception; Posture; Glenohumeral and scapulothoracic kinematics; Long term effects
MeSH Terms: conditions — Pain | interventions — TES

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Strenghtening + a-TES real (Experimental): Protocol of therapeutic exercises + real transcranial electrical stimulation of 8 weeks duration (24 supervised sessions). The program will consist of exercises to strengthen the RM and the scapulothoracic muscles, but the EG will perform the RM strengthening exercises while receiving real a-tDCS.
  Interventions: Other: Strenghtening + TES
- Strenghtening + a-TES placebo (Sham Comparator): Protocol of therapeutic exercises + placebo transcranial electrical stimulation of 8 weeks duration (24 supervised sessions). The program will consist of exercises to strengthen the RM and the scapulothoracic muscles, but the CG will perform the RM strengthening exercises while receiving placebo a-tDCS.
  Interventions: Other: Strenghtening + TES

INTERVENTIONS:
Other: Strenghtening + TES — Strenghtening of rotator cuff and scapulothoracic muscles protocol with the incorporation of anodal transcranial direct stimulation (real if experimental or sham if control)

SUMMARY:
The goal of this clinical trial is to analyze whether a physiotherapy protocol based on strengthening exercises to the shoulder girdle muscles carried on during anodal transcranial electrical stimulation (a-TES) is more effective on the symptoms and functionality of subjects with subacromial pain syndrome than an isolated strengthening program.

The main questions it aims to answer are:

* Is the strengthening + a-TES protocol effective on functionality?
* Is the strengthening + a-TES protocol effective on quality of life?
* Is the strengthening + a-TES protocol effective on pain?
* Is the strengthening + a-TES protocol effective on muscle strength?
* Is the strengthening + a-TES protocol effective on active range of movement?
* Is the strengthening + a-TES protocol effective on proprioception?
* Is the strengthening + a-TES protocol effective on posture?
* Is the strengthening + a-TES protocol effective on glenohumeral and scapulothoracic kinematics?

Participants will perform an 8 weeks-3 days/week shoulder strengthening protocol for the rotator cuff and scapulothoracic muscles using elastic bands and dumbbells. The rotator cuff exercises will be performed while they receive a-TES using a neoprene helmet with the electrodes placed in the opposite hemisphere to the affected side. The scapulothoracic exercises will be performed without the transcranial stimulation.

The experimental group will receive real a-TES, and will be compared with a control group that will perform the same therapeutic exercises but with placebo a-TES to see the effectiveness of the a-TES on the outcomes cited above.

DETAILED DESCRIPTION:
The project has obtained the approval of the Ethics Committee of the University of Valencia on June 6, 2023 (Id: UV-INV_ETICA-2701990).

The intervention will take place in the laboratories of the Physiotherapy Department of the University of Valencia. All the participants, once they have signed the informed consent and, after being randomly assigned to the EG or the CG, will be evaluated before starting the treatment (T0). A post-intervention evaluation will be carried one day after the end of the 24 sessions (T1), and a follow-up evaluation 3 weeks after the intervention (T2).

Subjects with unilateral shoulder pain will be recruited through social media and posters posted in primary care centers, hospitals, and other related locations.

The study will be triple blind: participants, evaluators and therapists. In order to monitor the possible adverse effects derived from the application of a-TES, the Bruitoni et al. Adverse Effects Questionnaire will be completed in each session. It is a questionnaire that contains 10 possible side effects (headache, neck pain, scalp pain, tingling, itching, burning, redness of the skin, drowsiness, concentration problems, severe mood change).If any of these symptoms occurred, the stimulation would be stopped and the next day would be tried again. If these effects were repeated, especially the headache or were of severe intensity, the patient would be withdrawn from the investigation.

The sample size has been calculated with the formula: n = (2 * (Zα/2 + Zβ) / d) ² (significance level of 0.05, Zα/2 = 1.96; Zβ =0.84, d= 0.5). Total, n= 64 subjects. In addition, the sample may be increased by 15% in anticipation of possible losses throughout the study (= 10 more subjects). Classic statistical methods will be used to calculate the mean as a measure of central tendency and the standard deviation as a measure of dispersion. Before carrying out the inferential analysis, the normal distribution of the sample will be checked using the Shapiro-Wilk test, homoscedasticity using the Levene test, and sphericity using the Mauchly test. Regarding the inferential analysis, a mixed ANOVA will be used with an intra-subject factor (time), with 4 categories, corresponding to the assessments made; and a between-subjects (group) factor corresponding to the assigned intervention. For post hoc comparisons, the Bonferroni adjustment will be used. In the event that the assumptions are not met, the corresponding non-parametric tests will be applied: Wilcoxon and Mann Whitney, adjusting the type I error. In the event of losses, the intention-to-treat procedure will be used for the statistical analysis of the data. .

ELIGIBILITY:
Subjects will be evaluated during a first consultation by a physiotherapist with experience in shoulder musculoskeletal pathology, following the algorithm for the diagnosis of shoulder problems, recommended by the British Elbow & Shoulder Society with the aim of detecting possible "flags red" and as a guide to rule out other shoulder pathologies that do not fit into the SDS. However, other tests will be added to ensure diagnostic accuracy, and these are described below.

Inclusion Criteria:

1. Age between 18 and 65 years.
2. Duration of pain greater than or equal to 3 months.
3. Presence of 3 or more of the following positive clinical tests:

   * painful arc
   * External rotation test against isometric resistance
   * Neer's test
   * Jobe test or empty can test
   * Hawkins-Kennedy test

Exclusion Criteria:

1. Previous shoulder or neck surgery.
2. History of shoulder fracture or dislocation.
3. Medical diagnosis of shoulder osteoarthritis.
4. Adhesive capsulitis
5. Cervicobrachialgia or reproducible shoulder pain with neck movements.
6. Clinical signs of total tear of the rotator cuff.
7. Corticosteroid injection in the previous 6 weeks.
8. Inflammatory disease, autoimmune or rheumatic, systemic (arthritis, lupus, myopathies).
9. Cognitive or behavioral problems that make it impossible to understand and follow the intervention (score less than 24 on the Mini-Mental State Examination Score) (73).
10. Any neurological or neoplastic disease.
11. Also those who present contraindications for transcranial electrical stimulation. For this, the recommendations of the checklist of Thair et al. which includes:

    * personal and family history of epilepsy
    * metal implants in the head
    * implanted medication pump
    * pacemaker
    * recurring headaches
    * skin diseases of the scalp (psoriasis, eczema)
    * head injuries
    * serious head surgeries
    * pregnancy
    * heart diseases
    * medications (psychotropics or antihistamines).

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Estimated)
Dates: Start 2023-11-23 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Changes in Pain and disability Index (SPADI), spanish version, scale. | Before the intervention, inmediately post intervention (and three months follow up.
  Scale for the measurement of Pain and disability related to shoulder disfunction. It contains 13 items, each with a score on a numerical scale from 0 (best) to 10 (worst). It consists of two domains: pain (of 5 items, score between 0-50) and disability (of 8 items, score between 0-80). In each domain the score can be expressed as a percentage. The total score of the scale is obtained as the sum of both domains (0 -100%). A higher score indicates greater pain-related disability.
Changes in Western Ontario Rotator cuff (WORC), spanish version, scale. | Before the intervention, inmediately post intervention (at eight weeks) and three months follow up.
  Scale for the measurement of the Quality of life related to shoulder disfunction. It consists of 21 questions, each with a visual analogue scale type response. The questions are grouped into 5 domains or sections: physical symptoms (6 items), sports and recreation (4 items), work (4 items), lifestyle (4 items) and emotions (3 items). Each item is measured on a 100 mm scale (from 0 best to 100 worst). So the worst value is 2100 and the best is 0.
Changes in a Visual Analogic scale, for the measurement of the shoulder intensity of pain | Before the intervention, inmediately post intervention (at eight weeks) and three months follow up.
  The intensity of the pain experienced in the affected shoulder at rest, at night and during activity in the last week will be evaluated. For this, a visual analogue scale (VAS) will be used. Subjects will mark pain intensity on a continuous horizontal line 10 cm long, labeled on the left end as "no pain" and on the right as "maximal pain".
Changes in shoulder pain pressure threshold (PPT) in Kg. | Before the intervention, inmediately post intervention (at eight weeks) and three months follow up.
  Mechanical sensitivity will be assessed using the Pressure Pain Threshold (PPT), which is defined as the minimum pressure at which the sensation of pressure changes to pain. The PPT will be measured with an analog algometer applied perpendicularly to the skin. The PPT will be evaluated on the affected side on: supraspinatus, infraspinatus, upper trapezius, levator scapulae, middle deltoid, C5-C6 interapophyseal joint and tibialis anterior. Higher PPT values (in Kg) will be interpreted as an improvement in mechanical sensitivity to pain in the tested areas.

SECONDARY OUTCOMES:
Changes in shoulder Muscle strenght measured by a dinamometer (Kg) | Before the intervention, inmediately post intervention (at eight weeks) and three months follow up.
  Shoulder strength will be quantified with a digital hand dynamometer for internal and external rotation, abduction, horizontal abduction, and scapular protraction on the affected side.
Changes in shoulder Active range of movement measured by goniometry (degrees) | Before the intervention, inmediately post intervention (at eight weeks) and three months follow up.
  A universal goniometer will be used to measure pain-free active range of motion of the affected shoulder for flexión, abduction and rotations.
Changes in Joint Position sense measured by the laser-pointer assisted angle reproduction (LP-ART), test (degrees). | Before the intervention, inmediately post intervention (at eight weeks) and three months follow up.
  A target with a central dot, drawn on a 1 x 1 m grid paper, will be placed 1 meter away the patient. The center of the target will be adjusted to the height of each participant and leveled horizontally to align with the glenohumeral joint, at the point where the assessor confirms 90° shoulder flexion-abduction using a goniometer.The evaluator will note the distance between both points (the target point and the point reached by the patient, in flexion and abduction) and the X and Y coordinates of the position reached with the pointer, in cm. With these data you will obtain the angular deviation of the target position
Changes in head forward posture, shoulder protraction and kiphosis (degrees) | Before the intervention, inmediately post intervention (at eight weeks) and three months follow up.
  For the head forward and shoulder protraction measurement, the participants will remain standing comfortably with their backs uncovered. Next, a photo of the cervicothoracic region will be taken with a digital camera. From the image, the angles will be measured, using ImageJ image measurement software.To measure dorsal kyphosis, two bubble inclinometers will be placed, one on T1 and T2 and the other on T12 and L1. The kyphosis angle will be the sum of both.
Changes in Subacromial space width measured by ultrasound (milimeters) | Before the intervention, inmediately post intervention (at eight weeks) and three months follow up.
  Distance between acromion and humerus head. The images will be captured with the participant seated in a chair, with the arm in three standardized positions: at 0˚, at 45˚ and at 60˚ of active abduction.
Changes in the scapulohumeral rithm (i.e., coordinated movement of the glenohumeral joint and the scapulothoracic joint) measured by al inclinometer (degrees). | Before the intervention, inmediately post intervention (at eight weeks) and three months follow up.
  The scapula measurement will be made at rest and during movement, at the moment the patient actively reaches the 60˚, 90˚ and 120˚ abduction positions. the glenohumeral-scapulothoracic ratio will be calculated in each position.
Changes in the mean signal amplitude of the scapulothoracic muscles measured by a surface electromiograph (µV) | Before the intervention, inmediately post intervention (at eight weeks) and three months follow up.
  Muscle activation of the Trapezius superior (TS), Trapezius inferior (TI), and anterior serratus (AS) will be measured at rest, at 60˚, 90˚, and 120˚ glenohumeral abduction. Each position will be held for 5 seconds. The surface electrodes will be placed according to the recommendations of the Surface Electromyography for the Non-Invasive Evaluation of Muscles (SENIAM) The mean signal amplitude (µV) will be calculated during the 5 seconds of muscle activation of the TS, TI and AS at each abduction angle.
Changes in the signal frequency of the scapulothoracic muscles measured by a surface electromiograph (Hz) | Before the intervention, inmediately post intervention (at eight weeks) and three months follow up.
  Muscle activation of the Trapezius superior (TS), Trapezius inferior (TI), and anterior serratus (AS) will be measured at rest, at 60˚, 90˚, and 120˚ glenohumeral abduction. Each position will be held for 5 seconds. The surface electrodes will be placed according to the recommendations of the Surface Electromyography for the Non-Invasive Evaluation of Muscles (SENIAM) The frequency will be calculated during the 5 seconds of muscle activation of the TS, TI and AS at each abduction angle.
Changes in the mean signal amplitud of primary motor cortex (M1) measured by EEG (µV) | Before and after each of the 24 sessions.
  The device (Starstim® tES-EEG systems, Neuroelectrics, Barcelona, Spain) will be used, with electrodes placed on the M1 motor area, connected to a neoprene helmet, to perform the electroencephalographic recording of cortical activity.The amplitude of the EEG peaks will be measured in µV.

CONTACTS AND LOCATIONS:
Locations (1):
- University of Valencia, Valencia, Valencia, Spain

IPD SHARING:
Plan to Share IPD: No